CLINICAL TRIAL: NCT00230373
Title: Evaluation of the Efficacy and Safety of Imiquimod 5% Cream in Plaque-type Morphea: A Pilot, Prospective Open-label Study
Brief Title: Imiquimod 5% Cream in Plaque-type Morphea: A Pilot, Prospective Open-label Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never started.
Sponsor: University of Alberta (Other)
Collaborators: 3M (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04CA05-IMIQ
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Morphea
Keywords: Localized scleroderma
MeSH Terms: conditions — Scleroderma, Localized | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: imiquimod 5% cream (Aldara)

SUMMARY:
Localized scleroderma or morphea is a fibrotic disease, imiquimod induces cytokines which inhibit fibrotic activity . We propose that topical imiquimod 5% cream is efficacious and safe in treating plaque-type morphea. Twenty adults will be enrolled for a pilot study. A screening and baseline clinic visit will be required for each patient enrolled in the study. Each visit will involve completing a medical history, skin examination, digital pictures, histologic examination if the patient consents and an ultrasonographic score. One morphea plaque will be treated with topical imiquimod 5% cream, and another morphea lesion with vehicle cream. Patients will be asked about side effects (local and systemic). Patients will be followed up in the clinic at 3, 6 and 9 months of therapy, and 3 months following end of treatment period (month 12).

ELIGIBILITY:
Inclusion Criteria:

* Adults and children > 6 years with plaque-type morphea
* Subject has not participated in previous study involving imiquimod for three months
* In the investigator's judgement, imiquimod treatment may benefit the patient over conventional treatment
* Subject has provided informed written consent
* Female subjects of childbearing potential have a pregnancy urine test that is negative prior to treatment
* Sexually active subjects agree to practice effective birth control throughout the duration of the study

Exclusion Criteria:

* Patients with a non-morphea skin disorder in the region of interest
* Subjects previously undergoing morphea therapy within four weeks of the study
* Subjects have a known hypersensitivity to imiquimod or component of the cream preparation
* Subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
The main outcome of this study is to evaluate the efficacy of imiquimod cream in improving morphea plaques. Improvement of skin induration will be measured by percent improvement in the skin induration as assessed radiologically by ultrasonography score.

SECONDARY OUTCOMES:
Any adverse outcome is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene T Dytoc, MD PhD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Dr. Marlene Dytoc's clinic, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Dr. Loretta Fiorillo's clinic, Red Deer, Alberta